CLINICAL TRIAL: NCT06683495
Title: Effect of Mirror Therapy on the Arteriovenous Fistula Cannulation-related Pain and Anxiety: A Prospective, Single Blind Randomized Controlled Study
Brief Title: Effect of Mirror Therapy on the Arteriovenous Fistula Cannulation-related Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Pain, Chronic; Fistula; Hemodialysis Complication
MeSH Terms: conditions — Chronic Pain; Fistula | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy (Experimental): For mirror therapy, a 50×40 cm mirror will be used. The patient will be positioned in a semi-sitting position at a 45° angle in bed, with the mirror placed on the side of the body where the access will be made. The arm with the fistula will be positioned behind the mirror. The position will be standardized so that the patient's thumb is 30 cm away from the mirror. The arm without the fistula will be supported with a pillow underneath to facilitate the patient's view in the mirror, positioned next to the patient. After observing their arm in the mirror for 15 minutes, the cannulation procedure will be performed.
  Interventions: Other: Mirror Therapy
- Routine Therapy (No Intervention): The routine procedure was performed. The fistula puncture was performed by the same nurse throughout the study.

INTERVENTIONS:
Other: Mirror Therapy — For mirror therapy, a 50×40 cm mirror will be used
  Arms: Mirror Therapy

SUMMARY:
Pharmacological and non-pharmacological methods are frequently used to reduce cannulation-related pain in patients with fistulas. Non-pharmacological approaches have been more favored than pharmacological approaches for some reasons, including ease of use and fewer side effects. Patients describe worry about the success of needling and resigned acceptance of pain and anxiety about dialysis needles. With this background in mind, mirror therapy has been introduced as one of the non-pharmacological interventions in the domain of pain management.

DETAILED DESCRIPTION:
Patients undergoing hemodialysis experience pain, anxiety and stress due to large-gauge needle punctures necessary to ensure efficient arteriovenous fistula flow. In addition, anxiety disorders are prevalent in hemodialysis patients, primarily caused by invasive procedures and dialysis machine alarm sounds. Patients describe worry about the success of needling and resigned acceptance of pain and anxiety about dialysis needles. Therefore, when performing an AVF puncture, nursing care should prioritise the management of pain and anxiety. With this background in mind, mirror therapy has been introduced as one of the non-pharmacological interventions in the domain of pain management. It has been reported that viewing the picture of a healthy limb could moderate pain perception in the affected one

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients who received hemodialysis (HD) treatment with an arteriovenous fistula (AVF) for at least 3 months
* Patients receiving HD treatment 3 days a week for 4 hours each session
* Patients with a pain score of ⩾1 during AVF cannulation, measured by a visual analog scale (VAS)
* Patients able to communicate in Turkish
* Patients without psychiatric disorders that impair communication
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients who were known to present difficulties with fistula cannulation (requiring multiple cannulations)
* Patients with a history of hematoma or stenosis in the arteriovenous fistula (AVF)
* Patients with an infection at the fistula site
* Patients who took painkillers within 3 hours prior to treatment
* Patients unable to maintain a sitting position on the bed
* Patients with low vision or visual disturbances (30 cm or less)
* Patients who did not wish to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Fistula Cannulation Related Pain | Up to 2 weeks (3 hemodialysis sessions in a week)
  It will be assessed six times at the end of the dialysis session with Visual Analogue Scale. Visual Analogue Scale ranging from 0 (no pain) to 10 (worst pain). Pain increases the score increases. The high point describes bad outcome
Change From Baseline Anxiety at Six Sessions | Up to 2 weeks ( 3 hemodialysis sessions in a week)
  It will be assessed with State-Trait Anxiety Inventory. This scale, which has a two-factor structure is comprised of 40 items. Twenty of these items assess the state anxiety status and the other 20 items assess trait anxiety. Each item is scored on a four-point scale. Total score ranges between 20 and 80 for anxiety. A high score indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Ozen, Assoc.Prof, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caglar S, Ozen N. Investigation of the effect of breathing exercise on invasive pain associated with arteriovenous fistula cannulation in hemodialysis patients: Randomized controlled, single-blind study. J Vasc Access. 2024 Nov;25(6):1940-1947. doi: 10.1177/11297298231194756. Epub 2023 Aug 24. PMID 37615173
- [Result] Alzaatreh MY, Abdalrahim MS. Management Strategies for Pain Associated with Arteriovenous Fistula Cannulation: An Integrative Literature Review. Hemodial Int. 2020 Jan;24(1):3-11. doi: 10.1111/hdi.12803. Epub 2019 Dec 3. PMID 31797508
- [Result] Ozen N, Tosun B, Sayilan AA, Eyileten T, Ozen V, Ecder T, Tosun N. Effect of the arterial needle bevel position on puncture pain and postremoval bleeding time in hemodialysis patients: A self-controlled, single-blind study. Hemodial Int. 2022 Oct;26(4):503-508. doi: 10.1111/hdi.13044. Epub 2022 Sep 6. PMID 36068183